CLINICAL TRIAL: NCT02440789
Title: Safety and Efficacy of Sirolimus for HIV Reservoir Reduction in Individuals on Suppressive Antiretroviral Therapy
Brief Title: Safety and Efficacy of Sirolimus for HIV Reservoir Reduction in Individuals on Suppressive Antiretroviral Therapy (ART)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5337; 2UM1AI068636 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-05-12 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2019-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Participants on a non-protease inhibitor (PI), non-non-nucleoside reverse transcriptase inhibitor (NNRTI) regimen, and for those on a non-PI, rilpivirine (RPV) based regimen received 0.025 mg/kg/day initial dose for 20 weeks.
  Participants on an NNRTI regimen with the exception of RPV received 0.05 mg/kg/day initial dose for 20 weeks.

SUMMARY:
The purpose of this study was to find out about the safety of sirolimus in individuals with HIV infection who were also being treated with ART. The investigators wanted to learn whether sirolimus decreases inflammation and immune activation in the body; whether sirolimus changes the level of HIV in the participants' blood; and how sirolimus interacts with ART in the blood. Sirolimus is approved by the Food and Drug Administration (FDA) to prevent organ rejection in patients aged 13 years and older receiving kidney transplants. Sirolimus had also been used for the prevention of complications after stem cell transplants and as a treatment for certain kinds of cancers in HIV-infected patients.

DETAILED DESCRIPTION:
The study was conducted with an initial lead-in period of 12 weeks where participants remained on ART, without study intervention. Samples were collected to define the pre-intervention steady-state of HIV, inflammation and immune activation parameters.

At week 12, sirolimus therapy was initiated for the planned 20 weeks of treatment. In order to achieve therapeutic levels, sirolimus therapy was initiated with lead-in dose of 0.025 or 0.05 mg/kg/day, depending on the ART regimen. Doses for each participant were then adjusted, based on trough blood sirolimus concentrations, to achieve target concentrations between 5 and 10 ng/mL. There were frequent initial visits for sirolimus trough concentration monitoring and potential dose adjustments, at weeks 12.5, 13, 13.5, 14, 14.5, 15, 15.5 and 16. Then visits occurred at weeks 18, 20, 24, 28 and 32. After the week 32 visit, the planned end of study treatment, there was an additional 12 weeks of post-sirolimus follow-up, with a final visit at week 44.

Study visits included physical examinations, clinical assessments, safety monitoring, and blood and oral swab collection. Anal swabs were collected at week 12 and 32. Samples were stored for subsequent protocol testing for the study outcomes.

In the primary analysis, the significance level was 0.05 for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On continuous ART for ≥24 months prior to study entry.
* CD4+ cell count ≥350 cells/mm^3
* Plasma HIV-1 RNA below the level of quantification for ≥24 months.
* White blood cell (WBC) ≥3000/mm^3
* Platelet count ≥125,000/mm^3
* Absolute neutrophil count (ANC) >1300/mm^3
* Aspartate aminotransferase (AST) <1.25 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) <1.25 x ULN
* Calculated creatinine clearance (CrCl) ≥60 mL/min
* Fasting or non-fasting triglyceride level ≤350 mg/dL
* Fasting or non-fasting LDL <160 mg/dL
* Urine protein to urine creatinine ratio ≤1 g/g from random urine collection

Exclusion Criteria:

* Serious illness requiring systemic treatment and/or hospitalization
* Documentation of any CDC Category C AIDS-indicator condition or oropharyngeal candidiasis (thrush)
* Intended modification of ART during the study.
* Latent tuberculosis (TB) infection
* TB disease within 48 weeks prior to study entry requiring treatment.
* History of active hepatitis B (HBV) infection.
* Hepatitis C virus (HCV) RNA-positive
* Previous myelodysplasia syndrome, lymphoproliferative disease, lung disease, malignancies, congestive heart failure, life-threatening fungal infection or herpes-zoster/varicella-zoster viral infection requiring treatment.
* Detectable Epstein-Barr virus (EBV) in blood
* Active infection other than HIV that required receipt of systemic antibiotic therapy by intravenous infusion
* History of major hypersensitivity reaction to macrolide drugs including angioedema, anaphylaxis, drug-induced dermatitis, or hypersensitivity vasculitis.
* Currently pregnant or breastfeeding, or planning to become pregnant prior to or during the study.
* Use of immunomodulators (eg, interleukins, interferons, and cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy.
* Active drug or alcohol use or dependence
* Vaccination within 14 days prior to study entry.
* On or planned to change to a PI-based ART or cobicistat-boosted regimen
* Anti-human papillomavirus (HPV) therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henrich, MD, Study Chair — University of California, San Francisco; Priscilla Hsue, MD, Study Chair — University of California, San Francisco
Locations (10):
- United States (10):
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Washington University CRS (2101), St Louis, Missouri
  - Weill Cornell Uptown CRS (7803), New York, New York
  - 31787 University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington

REFERENCES:
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.niaid.nih.gov/
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual) Version 2.0 January 2010 — https://rsc.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 10 Clinical Research Sites (CRSs) in the United States between December 2015 and March 2017.
Period: Overall Study
Arm/Group | Sirolimus
Started | 32
Initiated Sirolimus (2 participants withdrew consent prior to initiating Sirolimus) | 30
Completed 20 Weeks of Sirolimus (14 participants completed less than 20 weeks of Sirolimus) | 16
Completed | 28
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Not willing to adhere to reqs | 1

BASELINE CHARACTERISTICS:
Population: Participants who initiated Sirolimus
Groups:
- Sirolimus: Participants on a non-protease inhibitor (PI), non-non-nucleoside reverse transcriptase inhibitor (NNRTI) regimen, and for those on a non-PI, rilpivirine (RPV) based regimen received 0.025 mg/kg/day initial dose for 20 weeks.
  Participants on an NNRTI regimen with the exception of RPV received 0.05 mg/kg/day initial dose for 20 weeks.
  Sirolimus
Arm/Group | Sirolimus
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Safety Population | 52 [46 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 8
  Race/Ethnicity: Black Non-Hispanic | 18
  Race/Ethnicity: Hispanic | 3
  Race/Ethnicity: More than one race | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
CD4+ T-cell counts [Median (Inter-Quartile Range); unit: cells/mm^3] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
  cells/mm^3 | 818 [635 to 1031]
HIV-1 Gag-specific CD8+ T-cells by intracellular staining for interferon (IFN)-gamma [Median (Inter-Quartile Range); unit: %Gag-specific IFN-gamma+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific IFN-gamma+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.1 [0.05 to 0.14]
CD4+ T-cell-associated HIV-1 RNA [Median (Inter-Quartile Range); unit: log10(copies/10^6 CD4+ T-cells)] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus
  log10(copies/10^6 CD4+ T-cells)
    number analyzed (Participants) | 16
    (all) | 2.57 [2.19 to 3.13]
HIV-1 RNA by single-copy assay (SCA) [Count of Participants; unit: Participants] — Population: n = 16 participants completed 20 weeks of Sirolimus.
  Participants
    Study Entry: number analyzed (Participants) | 16
    Study Entry: < 0.7 copies/mL | 8
    Study Entry: >= 0.7 copies/mL | 8
    Study Week 12: number analyzed (Participants) | 16
    Study Week 12: < 0.7 copies/mL | 9
    Study Week 12: >= 0.7 copies/mL | 7
HIV-1 RNA [Count of Participants; unit: Participants] — Population: n = 16 participants completed 20 weeks of Sirolimus.
  Participants
    Study Entry: number analyzed (Participants) | 16
    Study Entry: < 40 copies/mL | 16
    Study Entry: >= 40 copies/mL | 0
    Study Week 12: number analyzed (Participants) | 16
    Study Week 12: < 40 copies/mL | 16
    Study Week 12: >= 40 copies/mL | 0
HIV-1 Gag-specific CD4+ T-cells by intracellular staining for IFN-gamma [Median (Inter-Quartile Range); unit: %Gag-specific IFN-gamma+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific IFN-gamma+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.04 [0.03 to 0.06]
GAG-specific CD107a+ CD8+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific CD107a+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific CD107a+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.01 [0 to 0.01]
GAG-specific CD107a+ CD4+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific CD107a+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific CD107a+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0 [0 to 0.01]
GAG-specific CD40L+ CD8+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific CD40L+CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific CD40L+CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.01 [0 to 0.03]
GAG-specific CD40L+ CD4+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific CD40L+CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific CD40L+CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.09 [0.05 to 0.12]
GAG-specific interleukin (IL)-2+ CD8+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific IL-2+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific IL-2+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.01 [0 to 0.03]
GAG-specific IL-2+ CD4+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific IL-2+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific IL-2+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.02 [0.01 to 0.03]
GAG-specific MIP1B+ CD8+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific MIP1B+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific MIP1B+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.06 [0.03 to 0.13]
GAG-specific MIP1B+ CD4+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific MIP1B+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific MIP1B+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.01 [0 to 0.01]
GAG-specific tumor necrosis factor (TNF)-alpha+ CD8+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific TNF-alpha CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific TNF-alpha CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.03 [0.02 to 0.05]
GAG-specific TNF-alpha+ CD4+ T-Cells [Median (Inter-Quartile Range); unit: %Gag-specific TNF-alpha CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Gag-specific TNF-alpha CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 0.03 [0.02 to 0.04]
%CD69+ CD4+ T-cells [Median (Inter-Quartile Range); unit: %CD69+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %CD69+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 5.5 [4.5 to 7.4]
%CD69+ CD8+ T-cells [Median (Inter-Quartile Range); unit: %CD69+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %CD69+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 8.4 [7.2 to 9.9]
%Ki67+ CD4+ T-cells [Median (Inter-Quartile Range); unit: %Ki67+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Ki67+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 2.2 [1.9 to 2.7]
%Ki67+ CD8+ T-cells [Median (Inter-Quartile Range); unit: %Ki67+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %Ki67+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 1.6 [1.4 to 1.8]
% programmed cell death protein 1 (PD1)+ CD4+ T-cells [Median (Inter-Quartile Range); unit: %PD1+ CD4+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %PD1+ CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 39.7 [31.3 to 42.6]
%PD1+ CD8+ T-cells [Median (Inter-Quartile Range); unit: %PD1+ CD8+ T-cells] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  %PD1+ CD8+ T-cells
    number analyzed (Participants) | 16
    (all) | 27.8 [21 to 39.3]
HIV-1 DNA levels in CD4+ T-cells [Median (Inter-Quartile Range); unit: log10(copies/10^6 CD4+ T-cells)] — Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12). Population: n = 16 participants completed 20 weeks of Sirolimus.
  log10(copies/10^6 CD4+ T-cells)
    number analyzed (Participants) | 16
    (all) | 2.72 [2.08 to 3.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met the Study-defined Composite Safety Endpoint
Description: The study-defined primary safety endpoint was a composite endpoint. A participant was considered to have met the endpoint if the participant 1) experienced a new Grade ≥3 Adverse Event (AE), including signs/symptoms, lab toxicity or clinical event, that was definitely, probably or possibly related to study treatment, as judged by the core team, or 2) had a change in CD4+ cell count ( confirmed >50% decline or to <300 cells/mm3) while on sirolimus. The screening visit occurred within 60 days of study entry.
Time Frame: Screening to study week 32 (week 20 of Sirolimus)
Population: Participants Initiating Sirolimus.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 30
Participants | 3

2. Primary Outcome: Efficacy - Immunologic: Frequency of HIV-1 Gag-specific CD8+ T-cells by Intracellular Staining for IFN-gamma
Description: Frequency of HIV-1 Gag-specific CD8+ T-cells by intracellular staining for IFN-gamma. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IFN-gamma+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific IFN-gamma+ CD8+ T-cells
  Baseline | 0.11 (0.08)
  Week 20 on Sirolimus: number analyzed (Participants) | 15
  Week 20 on Sirolimus | 0.11 (0.07)

3. Primary Outcome: Efficacy - Immunologic: Change in HIV-1 Gag-specific CD8+ T-cells by Intracellular Staining for IFN-gamma
Description: Change in HIV-1 Gag-specific CD8+ T-cells by intracellular staining for IFN-gamma (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IFN-gamma+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific IFN-gamma+ CD8+ T-cells | -0.01 (0.06)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.56, t-test, 2 sided; paired t-test

4. Primary Outcome: Efficacy - Virologic: CD4+ T-cell-associated HIV-1 RNA
Description: CD4+ T-cell-associated HIV-1 RNA. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: log10(copies/10^6 CD4+ T-cells)
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
log10(copies/10^6 CD4+ T-cells)
  Baseline | 2.56 (0.67)
  Week 20 on Sirolimus | 2.35 (0.68)

5. Primary Outcome: Efficacy - Virologic: Change in CD4+ T-cell-associated HIV-1 RNA
Description: Change in CD4+ T-cell-associated HIV-1 RNA (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: log10(copies/10^6 CD4+ T-cells)
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
log10(copies/10^6 CD4+ T-cells) | -0.21 (0.48)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.11, t-test, 2 sided; paired t-test

6. Primary Outcome: Efficacy - Virologic: Plasma HIV-1 RNA by SCA
Description: Plasma HIV-1 RNA by SCA
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
Participants
  Study week 0: < 0.7 copies/mL | 8
  Study week 0: >= 0.7 copies/mL | 8
  Study week 12: < 0.7 copies/mL | 9
  Study week 12: >= 0.7 copies/mL | 7
  Study week 32 (week 20 on Sirolimus): < 0.7 copies/mL | 8
  Study week 32 (week 20 on Sirolimus): >= 0.7 copies/mL | 8

7. Primary Outcome: Efficacy - Virologic: Change in Plasma HIV-1 RNA by SCA
Description: Change in plasma HIV-1 RNA by SCA (week 32 measurement minus baseline measurement).
  Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: log10(copies/mL)
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
log10(copies/mL) | -0.01 (0.47)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.93, t-test, 2 sided; paired t-test; results less than the analysis lower limit (0.7 cp/mL) were imputed to a value of one half the analysis lower limit

8. Secondary Outcome: Measurement of CD4+ T-cell Counts
Description: CD4+ T-cell counts. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
cells/mm^3
  Baseline | 937 (402)
  Study week 16 (week 4 on Sirolimus) | 858 (403)
  Study week 24 (week 12 on Sirolimus) | 820 (378)
  Study week 32 (week 20 on Sirolimus) | 820 (377)
  Study week 44 | 891 (320)

9. Secondary Outcome: Change in CD4+ T-cell Counts
Description: Change in CD4+ T-cell counts (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
cells/mm^3 | -118 (211)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.041, t-test, 2 sided; paired t-test

10. Secondary Outcome: Measurement of HIV-1 RNA Levels
Description: HIV-1 RNA levels by conventional assay
Time Frame: weeks 0, 12, (pre-Sirolimus) 16, 24, 32 (4, 12, 20 weeks on Sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
Participants
  Study Week 0: < 40 copies/mL | 16
  Study Week 0: >= 40 copies/mL | 0
  Study Week 12: < 40 copies/mL | 16
  Study Week 12: >= 40 copies/mL | 0
  Study Week 16 (Week 4 on Sirolimus): < 40 copies/mL | 16
  Study Week 16 (Week 4 on Sirolimus): >= 40 copies/mL | 0
  Study Week 24 (Week 12 on Sirolimus): < 40 copies/mL | 16
  Study Week 24 (Week 12 on Sirolimus): >= 40 copies/mL | 0
  Study Week 32 (Week 20 on Sirolimus): < 40 copies/mL | 16
  Study Week 32 (Week 20 on Sirolimus): >= 40 copies/mL | 0
  Study Week 44: < 40 copies/mL | 16
  Study Week 44: >= 40 copies/mL | 0

11. Secondary Outcome: Cell-associated HIV-1 DNA Levels in Total CD4+ Cells
Description: HIV-1 DNA levels in CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: log10(copies/10^6 CD4+ T-cells)
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
log10(copies/10^6 CD4+ T-cells)
  Baseline | 2.65 (0.71)
  Study week 16 (week 4 on Sirolimus) | 2.45 (0.81)
  Study week 24 (week 12 on Sirolimus) | 2.48 (0.78)
  Study week 32 (week 20 on Sirolimus) | 2.49 (0.75)
  Study week 44 | 2.51 (0.79)

12. Secondary Outcome: Change in Cell-associated HIV-1 DNA Levels in Total CD4+ Cells
Description: Change in HIV-1 DNA levels in CD4+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: log10(copies/10^6 CD4+ T-cells)
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
log10(copies/10^6 CD4+ T-cells) | -0.16 (0.21)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.008, t-test, 2 sided; paired t-test

13. Secondary Outcome: Measurement of HIV-1 Gag-specific CD107a+ CD8+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific CD107a+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific CD107a+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Gag-specific CD107a+ CD8+ T-cells
  Baseline | 0.01 (0.01)
  Study week 16 (week 4 on Sirolimus) | 0.02 (0.02)
  Study week 24 (week 12 on Sirolimus) | 0.01 (0.01)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.05 (0.14)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.02 (0.03)

14. Secondary Outcome: Change in HIV-1 Gag-specific CD107a+ CD8+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific CD107a+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific CD107a+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%Gag-specific CD107a+ CD8+ T-cells | 0.04 (0.14)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.26, t-test, 2 sided; paired t-test

15. Secondary Outcome: Measurement of HIV-1 Gag-specific CD40L+ CD8+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific CD40L+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific CD40L+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Gag-specific CD40L+ CD8+ T-cells
  Baseline | 0.02 (0.02)
  Study week 16 (week 4 on Sirolimus) | 1.15 (4.53)
  Study week 24 (week 12 on Sirolimus) | 0.01 (0.03)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.03 (0.05)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.01 (0.02)

16. Secondary Outcome: Change in HIV-1 Gag-specific CD40L+ CD8+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific CD40L+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific CD40L+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%Gag-specific CD40L+ CD8+ T-cells | 0.01 (0.06)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.75, t-test, 2 sided; paired t-test

17. Secondary Outcome: Measurement of HIV-1 Gag-specific IL-2+ CD8+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific IL-2+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific IL-2+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Gag-specific IL-2+ CD8+ T-cells
  Baseline | 0.02 (0.03)
  Study week 16 (week 4 on Sirolimus) | 0.01 (0.02)
  Study week 24 (week 12 on Sirolimus) | 0.02 (0.02)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.02 (0.03)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.03 (0.04)

18. Secondary Outcome: Change in HIV-1 Gag-specific IL-2+ CD8+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific IL-2+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Gag-specific IL-2+ CD8+ T-cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%Gag-specific IL-2+ CD8+ T-cells | 0 (0.05)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.97, t-test, 2 sided; paired t-test

19. Secondary Outcome: Measurement of HIV-1 Gag-specific MIP1B+ CD8+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific MIP1B+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific MIP1B+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific MIP1B+ CD8+ T-Cells
  Baseline | 0.09 (0.08)
  Study week 16 (week 4 on Sirolimus) | 0.51 (1.72)
  Study week 24 (week 12 on Sirolimus) | 0.08 (0.08)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.09 (0.08)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.08 (0.1)

20. Secondary Outcome: Change in HIV-1 Gag-specific MIP1B+ CD8+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific MIP1B+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific MIP1B+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific MIP1B+ CD8+ T-Cells | -0.01 (0.06)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.7, t-test, 2 sided; paired t-test

21. Secondary Outcome: Measurement of HIV-1 Gag-specific TNF-alpha+ CD8+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific TNF-alpha+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific TNF-a+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific TNF-a+ CD8+ T-Cells
  Baseline | 0.04 (0.03)
  Study week 16 (week 4 on Sirolimus) | 0.04 (0.03)
  Study week 24 (week 12 on Sirolimus) | 0.03 (0.02)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.05 (0.05)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.04 (0.04)

22. Secondary Outcome: Change in HIV-1 Gag-specific TNF-alpha+ CD8+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific TNF-alpha+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific TNF-a+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific TNF-a+ CD8+ T-Cells | 0.01 (0.04)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.47, t-test, 2 sided; paired t-test

23. Secondary Outcome: Measurement of HIV-1 Gag-specific CD4+ T-cell by Intracellular Staining for IFN-gamma Responses
Description: Frequency of HIV-1 Gag-specific CD4+ T-cells by intracellular staining for IFN-gamma. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IFN-g+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific IFN-g+ CD4+ T-Cells
  Baseline | 0.06 (0.06)
  Study week 16 (week 4 on Sirolimus) | 0.04 (0.03)
  Study week 24 (week 12 on Sirolimus) | 0.05 (0.06)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.06 (0.05)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.04 (0.04)

24. Secondary Outcome: Change in HIV-1 Gag-specific CD4+ T-cell by Intracellular Staining for IFN-gamma Responses
Description: Change in HIV-1 Gag-specific CD4+ T-cells by intracellular staining for IFN-gamma (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IFN-g+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific IFN-g+ CD4+ T-Cells | 0 (0.04)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.72, t-test, 2 sided; paired t-test

25. Secondary Outcome: Measurement of HIV-1 Gag-specific CD107a+ CD4+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific CD107a+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific CD107a+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific CD107a+ CD4+ T-Cells
  Baseline | 0.01 (0.01)
  Study week 16 (week 4 on Sirolimus) | 0.01 (0.01)
  Study week 24 (week 12 on Sirolimus) | 0.01 (0.01)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.03 (0.08)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.02 (0.02)

26. Secondary Outcome: Change in HIV-1 Gag-specific CD107a+ CD4+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific CD107a+ CD4+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific CD107a+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific CD107a+ CD4+ T-Cells | 0.02 (0.08)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.28, t-test, 2 sided; paired t-test

27. Secondary Outcome: Measurement of HIV-1 Gag-specific CD40L+ CD4+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific CD40L+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific CD40L+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific CD40L+ CD4+ T-Cells
  Baseline | 0.08 (0.05)
  Study week 16 (week 4 on Sirolimus) | 0.06 (0.06)
  Study week 24 (week 12 on Sirolimus) | 0.1 (0.06)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.08 (0.07)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.08 (0.07)

28. Secondary Outcome: Change in HIV-1 Gag-specific CD40L+ CD4+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific CD40L+ CD4+ T-cells (week 32 measurement minus baseline measurement).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific CD40L+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific CD40L+ CD4+ T-Cells | -0.01 (0.07)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.7, t-test, 2 sided; paired t-test

29. Secondary Outcome: Measurement of HIV-1 Gag-specific IL-2+ CD4+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific IL-2+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IL-2+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific IL-2+ CD4+ T-Cells
  Baseline | 0.03 (0.05)
  Study week 16 (week 4 on Sirolimus) | 0.04 (0.03)
  Study week 24 (week 12 on Sirolimus) | 0.04 (0.07)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.08 (0.16)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.04 (0.05)

30. Secondary Outcome: Change in HIV-1 Gag-specific IL-2+ CD4+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific IL-2+ CD4+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific IL-2+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific IL-2+ CD4+ T-Cells | 0.04 (0.15)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.28, t-test, 2 sided; paired t-test

31. Secondary Outcome: Measurement of HIV-1 Gag-specific MIP1B+ CD4+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific MIP1B+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific MIP1B+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific MIP1B+ CD4+ T-Cells
  Baseline | 0.01 (0.01)
  Study week 16 (week 4 on Sirolimus) | 0.01 (0.01)
  Study week 24 (week 12 on Sirolimus) | 0.01 (0.02)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.01 (0.01)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.01 (0.01)

32. Secondary Outcome: Change in HIV-1 Gag-specific MIP1B+ CD4+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific MIP1B+ CD4+ T-cells (week 32 measurement minus baseline measurement).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific MIP1B+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific MIP1B+ CD4+ T-Cells | 0 (0.01)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.77, t-test, 2 sided; paired t-test

33. Secondary Outcome: Measurement of HIV-1 Gag-specific TNF-alpha+ CD4+ T-cell Responses
Description: Frequency of HIV-1 Gag-specific TNF-alpha+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific TNF-alpha+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%GAG-specific TNF-alpha+ CD4+ T-Cells
  Baseline | 0.04 (0.03)
  Study week 16 (week 4 on Sirolimus) | 0.04 (0.03)
  Study week 24 (week 12 on Sirolimus) | 0.03 (0.04)
  Study week 32 (week 20 on Sirolimus): number analyzed (Participants) | 15
  Study week 32 (week 20 on Sirolimus) | 0.04 (0.03)
  Study week 44: number analyzed (Participants) | 15
  Study week 44 | 0.04 (0.03)

34. Secondary Outcome: Change in HIV-1 Gag-specific TNF-alpha+ CD4+ T-cell Responses
Description: Change in frequency of HIV-1 Gag-specific TNF-alpha+ CD4+ T-cells (week 32 measurement minus baseline measurement).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %GAG-specific TNF-alpha+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 15
%GAG-specific TNF-alpha+ CD4+ T-Cells | 0 (0.02)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.93, t-test, 2 sided; paired t-test

35. Secondary Outcome: Measurement of %CD69+ CD4+ T-cells
Description: Measurement of %CD69+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %CD69+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%CD69+ CD4+ T-Cells
  Baseline | 6.3 (2.6)
  Study week 16 (week 4 on Sirolimus) | 6.1 (2.3)
  Study week 24 (week 12 on Sirolimus) | 5.8 (2.0)
  Study week 32 (week 20 on Sirolimus) | 6.1 (1.9)
  Study week 44 | 5.9 (2.3)

36. Secondary Outcome: Change in of %CD69+ CD4+ T-cells
Description: Change in of %CD69+ CD4+ T-cells (week 32 measurement minus baseline measurement).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %CD69+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%CD69+ CD4+ T-Cells | -0.17 (1.51)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.65, t-test, 2 sided; paired t-test

37. Secondary Outcome: Measurement of %CD69+ CD8+ T-cells
Description: Measurement of %CD69+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %CD69+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%CD69+ CD8+ T-Cells
  Baseline | 8.6 (2.9)
  Study week 16 (week 4 on Sirolimus) | 8.4 (2.8)
  Study week 24 (week 12 on Sirolimus) | 7.9 (2.5)
  Study week 32 (week 20 on Sirolimus) | 8.1 (2.5)
  Study week 44 | 8.2 (2.4)

38. Secondary Outcome: Change in of %CD69+ CD8+ T-cells
Description: Change in of %CD69+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %CD69+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%CD69+ CD8+ T-Cells | -0.52 (1.63)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.22, t-test, 2 sided; paired t-test

39. Secondary Outcome: Measurement of %Ki67+ CD4+ T-cells
Description: Measurement of %Ki67+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Ki67+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Ki67+ CD4+ T-Cells
  Baseline | 2.4 (0.8)
  Study week 16 (week 4 on Sirolimus) | 2.2 (0.9)
  Study week 24 (week 12 on Sirolimus) | 2.2 (0.8)
  Study week 32 (week 20 on Sirolimus) | 1.9 (0.8)
  Study week 44 | 2.4 (1)

40. Secondary Outcome: Change in of %Ki67+ CD4+ T-cells
Description: Change in of %Ki67+ CD4+ T-cells (week 32 measurement minus baseline measurement).
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Ki67+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Ki67+ CD4+ T-Cells | -0.51 (0.86)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.031, t-test, 2 sided; paired t-test

41. Secondary Outcome: Measurement of %Ki67+ CD8+ T-cells
Description: Measurement of %Ki67+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Ki67+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Ki67+ CD8+ T-Cells
  Baseline | 1.8 (0.8)
  Study week 16 (week 4 on Sirolimus) | 1 (0.4)
  Study week 24 (week 12 on Sirolimus) | 1.4 (0.7)
  Study week 32 (week 20 on Sirolimus) | 1.2 (0.6)
  Study week 44 | 1.7 (0.7)

42. Secondary Outcome: Change in of %Ki67+ CD8+ T-cells
Description: Change in of %Ki67+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %Ki67+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%Ki67+ CD8+ T-Cells | -0.54 (0.67)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.005, t-test, 2 sided; paired t-test

43. Secondary Outcome: Measurement of %PD1+ CD4+ T-cells
Description: Measurement of %PD1+ CD4+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %PD1+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%PD1+ CD4+ T-Cells
  Baseline | 38.4 (9.6)
  Study week 16 (week 4 on Sirolimus) | 39 (11.1)
  Study week 24 (week 12 on Sirolimus) | 38.8 (10.7)
  Study week 32 (week 20 on Sirolimus) | 38.8 (9.9)
  Study week 44 | 35.5 (10.6)

44. Secondary Outcome: Change in of %PD1+ CD4+ T-cells
Description: Change in of %PD1+ CD4+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %PD1+ CD4+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%PD1+ CD4+ T-Cells | 0.42 (4.19)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.69, t-test, 2 sided; paired t-test

45. Secondary Outcome: Measurement of %PD1+ CD8+ T-cells
Description: Measurement of %PD1+ CD8+ T-cells. Baseline is the mean of the two pre-Sirolimus measurements (study entry and study week 12).
Time Frame: At study weeks 0, 12, 16, 24, 32 (4, 12, 20 weeks on sirolimus) and 44
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %PD1+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%PD1+ CD8+ T-Cells
  Baseline | 29.4 (10.2)
  Study week 16 (week 4 on Sirolimus) | 28.4 (9.9)
  Study week 24 (week 12 on Sirolimus) | 28.4 (10.6)
  Study week 32 (week 20 on Sirolimus) | 26.6 (9.9)
  Study week 44 | 25.5 (8.7)

46. Secondary Outcome: Change in of %PD1+ CD8+ T-cells
Description: Change in of %PD1+ CD8+ T-cells (week 32 measurement minus baseline measurement)
Time Frame: At study weeks 0, 12 and 32 (week 20 on Sirolimus)
Population: Participants completing 20 weeks of Sirolimus
Measure: Mean (Standard Deviation); unit: %PD1+ CD8+ T-Cells
Arm/Group | Sirolimus
Number analyzed (Participants) | 16
%PD1+ CD8+ T-Cells | -2.85 (3.74)
Statistical Analysis 1: Comparison: Sirolimus; Test type: Other; p = 0.008, t-test, 2 sided; paired t-test

ADVERSE EVENTS:
Time Frame: Screening to study week 32 (week 20 of Sirolimus)
Description: At entry, all grades of signs and symptoms that occurred within 30 days before entry were recorded; post-entry, all grades of Grade ≥2 were recorded. All Grade 3 or higher sign/symptom, any sign/symptom regardless of grade that led to a change in study treatment, or that met ICH, EAE or SAE guidelines were recorded. The DAIDS AE Grading Table Version 2.0 and Expedited AE Manual Version 2.0 were used.
  All participants exposed to Sirolimus are included.
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=30)
Diarrhoea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=30)
Diarrhoea (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 3
Malaise (General disorders) | 3
Pain (General disorders) | 3
Pyrexia (General disorders) | 2
Viral upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 15
Blood creatine phosphokinase increased (Investigations) | 5
Blood creatinine increased (Investigations) | 3
Blood glucose decreased (Investigations) | 3
Blood glucose increased (Investigations) | 13
Blood pressure increased (Investigations) | 2
Blood sodium decreased (Investigations) | 3
Blood sodium increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 18
Low density lipoprotein increased (Investigations) | 13
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT02440789/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT02440789/SAP_000.pdf